CLINICAL TRIAL: NCT03283930
Title: A Clinical Trial of a Gamified Attention Bias Modification Training in Anxious Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0192A
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-11

CONDITIONS: Anxiety Disorders
Keywords: Cognitive Behavioral Therapy (CBT); Attention; Anxiety; Children; Adolescents
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients with anxiety disorders are assessed on a number of mental health and biological variables. Patients who can agree to attend regular psychotherapy sessions are randomized to receive cognitive behavioral therapy with computer-based augmentation. In one study arm, these patients receive cognitive behavioral therapy with an active form of a computer game. In the other treatment arm, subjects receive cognitive behavioral therapy with a control treatment.
Who Masked: Participant, Investigator
Masking Description: The active and control treatment arms differ in the spatial arrangements of figures on a computer screen. Because these figures are presented for very brief periods of time, subjects cannot easily decipher differences in the arrangements across the active and control treatments. All study team members who work with patients remain blind to the treatment conditions as well.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Experimental): Children and adolescent participants with anxiety disorder receive cognitive behavioral therapy (CBT) for a 12-week period. In the final eight weeks of the trial, the subjects complete the Active Attention Bias Modification Training (ABMT), computer-based attention bias modification training aimed at re-training attentional biases before a CBT session: Part 1. modified dot-probe task, where a target is always presented at the previous location of the neutral and not the simultaneously presented threatening stimulus. Part 2. visual search, where the targets are always presented distally of threatening distractors.
  Interventions: Behavioral: Active Attention Bias Modification Training
- Control Intervention (Placebo Comparator): Children and adolescent participants with anxiety disorder receive cognitive behavioral therapy (CBT) for a 12-week period. In the final eight weeks of the trial, the subjects complete the control intervention before a CBT session: Part 1. dot-probe task, where a target is equally randomly presented at the previous location of the neutral or the simultaneously presented threatening stimulus. Part 2. visual search, where the targets are equally randomly presented distal of neutral and threatening distractors.
  Interventions: Behavioral: Placebo Attention Bias Modification Training

INTERVENTIONS:
Behavioral: Active Attention Bias Modification Training — Computer-based attention bias modification training administered at weekly CBT session aimed at re-training attentional biases
  Arms: Active Intervention
Behavioral: Placebo Attention Bias Modification Training
  Arms: Control Intervention

SUMMARY:
Background: Attention bias modification training (ABMT) and cognitive behavioral therapy (CBT) likely target different aspects of aberrant threat responses in anxiety disorders and may be combined to maximize therapeutic benefit. However, studies investigating the effect of ABMT in the context of CBT have yielded mixed results.

Objective: The primary goal of this project is to utilize an enhanced ABMT to target attentional bias towards threat, in addition to classic CBT for anxiety disorders in youth, to determine the efficacy of ABMT in the context of CBT.

Study Population: 121 youth (8-17 years old) with a primary anxiety disorder diagnosis

Methods: In this sub-study,

* Participants will receive open CBT treatment.
* Open CBT treatment will be augmented with computer-based attention retraining, delivered in a randomized-controlled design, with random assignment to either active or placebo attention-training regimens.
* This enhanced ABMT integrates a modified dot-probe task used in previous studies, where a target is always presented at the previous location of the neutral and not the simultaneously presented threatening stimulus, with a visual search, where the targets are always presented distally of threatening distractors.
* These two training elements (modified dot-probe and visual search) will be embedded in an engaging game to foster motivation and adherence.

Outcome: Symptom improvement will be compared between the two study arms.

DETAILED DESCRIPTION:
Background: Attention bias modification training (ABMT) and cognitive behavioral therapy (CBT) likely target different aspects of aberrant threat responses in anxiety disorders and may be combined to maximize therapeutic benefit. However, studies investigating the effect of ABMT in the context of CBT have yielded mixed results.

Objective: The primary goal of this project is to utilize an enhanced ABMT to target attentional bias towards threat, in addition to classic CBT for anxiety disorders in youth, to determine the efficacy of ABMT in the context of CBT.

Study Population: 121 youth (8-17 years old) with a primary anxiety disorder diagnosis who are originally consented on 01-M-0192 will be recruited and randomized to each arm in the sub-study

Methods: In this sub-study,

* Participants will receive open CBT treatment.
* Open CBT treatment will be augmented with computer-based attention retraining, delivered in a randomized-controlled design, with random assignment to either active or placebo attention-training regimens.
* This enhanced ABMT integrates a modified dot-probe task used in previous studies, where a target is always presented at the previous location of the neutral and not the simultaneously presented threatening stimulus, with a visual search, where the targets are always presented distally of threatening distractors.
* These two training elements (modified dot-probe and visual search) will be embedded in an engaging game to foster motivation and adherence.

Outcome: Symptom improvement will be compared between the two study arms at different times using

* The Pediatric Anxiety Rating Scale (PARS)
* The Clinical Global Impression of Improvement Scale (CGI-I)
* The Children's Global Assessment Scale (CGAS)
* The Screen for Child Anxiety Related Disorders (SCARED)
* The State-Trait Anxiety Inventory for Children (STAI-C)
* The Self-Efficacy Questionnaire (SEQ-C)

ELIGIBILITY:
INCLUSION CRITERIA:

-ALL JUVENILE SUBJECTS WITH AN ANXIETY DISORDER:

* Diagnosis: Current Diagnosis of Social Phobia, Separation Anxiety, Generalized Anxiety Disorder, or Panic Disorder (Based on K-SADS (juveniles))
* Symptom Severity: Clinically significant, ongoing anxiety symptoms
* Clinical Impairment: Clinically significant, ongoing distress or impairment from anxiety
* Age: 8 - 17 (subjects who consent as 17- year-olds but turn 18 during the course of the study will be eligible to complete all procedures completed by other subjects who consent as 17- year- old but do not turn 18).
* Consent: can give consent/assent (Parents will provide consent; minors will provide assent)
* IQ: all subjects will have intelligence quotient (IQ) > 70 (Assessment relies on WASI)
* Language: all subjects will speak English

EXCLUSION CRITERIA:

* Any serious medical condition or condition that interferes with participation
* Pregnancy
* Current use of any psychoactive substance; current suicidal ideation; current diagnosis of attention deficit hyperactivity disorder (ADHD) of sufficient severity to require pharmacotherapy.
* Current diagnoses Tourette's Disorder, obsessive compulsive disorder (OCD), post-traumatic distress disorder, conduct disorder
* Past or current history of mania, psychosis, or severe pervasive developmental disorder
* Recent use of an selective serotonin reuptake inhibitor (SSRI); all subjects must have been free of any SSRI-use for at least one month (fluoxetine six months) and must not have been treated with an SSRI for their current depressive episode.
* National Institute of Mental Health (NIMH) employees and staff and their immediate family members will be excluded from the study per NIMH policy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- NIH Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Britton JC, Suway JG, Clementi MA, Fox NA, Pine DS, Bar-Haim Y. Neural changes with attention bias modification for anxiety: a randomized trial. Soc Cogn Affect Neurosci. 2015 Jul;10(7):913-20. doi: 10.1093/scan/nsu141. Epub 2014 Oct 24. PMID 25344944
- [Background] White LK, Sequeira S, Britton JC, Brotman MA, Gold AL, Berman E, Towbin K, Abend R, Fox NA, Bar-Haim Y, Leibenluft E, Pine DS. Complementary Features of Attention Bias Modification Therapy and Cognitive-Behavioral Therapy in Pediatric Anxiety Disorders. Am J Psychiatry. 2017 Aug 1;174(8):775-784. doi: 10.1176/appi.ajp.2017.16070847. Epub 2017 Apr 14. PMID 28407726
- [Background] Linke JO, Jones E, Pagliaccio D, Swetlitz C, Lewis KM, Silverman WK, Bar-Haim Y, Pine DS, Brotman MA. Efficacy and mechanisms underlying a gamified attention bias modification training in anxious youth: protocol for a randomized controlled trial. BMC Psychiatry. 2019 Aug 7;19(1):246. doi: 10.1186/s12888-019-2224-2. PMID 31391027
- [Derived] Byrne ME, Haller SP, Linke JO, Lewis KM, Berman ED, Henry LM, Pagliaccio D, Quezada D, Meyer M, Abend R, Kircanski K, Silverman WK, Lazarov A, Bar-Haim Y, Brotman MA, Pine DS. Gamified Attention Bias Modification Training to Augment Cognitive-Behavioral Therapy for Youth Anxiety Disorders: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2025 Aug 22:S0890-8567(25)01428-5. doi: 10.1016/j.jaac.2025.08.010. Online ahead of print. PMID 40850530
- [Derived] Lewis KM, Matsumoto C, Cardinale E, Jones EL, Gold AL, Stringaris A, Leibenluft E, Pine DS, Brotman MA. Self-Efficacy As a Target for Neuroscience Research on Moderators of Treatment Outcomes in Pediatric Anxiety. J Child Adolesc Psychopharmacol. 2020 May;30(4):205-214. doi: 10.1089/cap.2019.0130. Epub 2020 Mar 11. PMID 32167803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Intervention | Control Intervention
Started | 59 | 62
Completed | 48 | 49
Not Completed | 11 | 13
Not completed — Scheduling conflict | 8 | 10
Not completed — Due to coronavirus disease 2019 (COVID-19) pandemic | 1 | 1
Not completed — Technical software issue | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Intervention | Control Intervention | Total
Number analyzed (Participants) | 59 | 62 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 62 | 121
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 23 | 25 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 47 | 54 | 101
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 41 | 46 | 87
  More than one race | 11 | 10 | 21
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Anxiety Rating Scale
Description: The Pediatric Anxiety Rating Scale (PARS) measures anxiety symptoms and related functional impairment in youth as continuous outcome. It comprises a 50- item checklist asking for seven dimensions of global severity/ impairment: Each item is rated on a 0- 5 scale by a clinician based on parent- and child-report. The sum score is calculated based on 5 of the 7 sub-scales and ranges from 0 to 25 with higher scores reflecting greater levels of anxiety. PARS score was measured at different time points during the study.
Time Frame: Weeks 3, 8, and 12
Population: The analyses included participants who were randomized to either arm of the study and had data available for analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Intervention | Control Intervention
Number analyzed (Participants) | 57 | 61
units on a scale
  Week 3 | 13.596491 (0.5472) | 14.557377 (0.4867)
  Week 8: number analyzed (Participants) | 56 | 58
  Week 8 | 11.50 (0.5500) | 12.206897 (0.5146)
  Week 12: number analyzed (Participants) | 57 | 55
  Week 12 | 9.666667 (0.66431) | 9.890909 (0.5564)

2. Primary Outcome: Clinical Global Impression of Improvement Scale
Description: The Clinical Global Impression of Improvement (CGI-I) scale is a measure of global symptom improvement rated by clinicians. Scores range from 1-7, with lower scores reflecting greater levels of improvement. This scale provides an ordinal outcome, as participants with CGI-I ratings less than or equal to 3 at week 8 are considered "responders" and participants with scores >3 at week 8 are considered "non-responders".
Time Frame: Week 8
Population: The analyses included participants who were randomized to either arm of the study and had data available for analysis.
Measure: Number; unit: participants
Arm/Group | Active Intervention | Control Intervention
Number analyzed (Participants) | 50 | 57
participants
  Responders | 11 | 16
  Non-Responders | 39 | 41

3. Secondary Outcome: Children's Global Assessment Scale
Description: The Children's Global Assessment Scale (CGAS) is a clinician-rated measure of global functioning, with scores ranging from 1 to 100. Higher score indicates better overall functioning.
Time Frame: Weeks 3, 8, and 12
Population: The analyses included participants who were randomized to either arm of the study and had data available for analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Intervention | Control Intervention
Number analyzed (Participants) | 57 | 57
units on a scale
  Week 3 | 54.38596 (0.9155282) | 54.38596 (0.9748576)
  Week 8: number analyzed (Participants) | 54 | 56
  Week 8 | 61.03704 (0.9076748) | 59.75000 (0.8083372)
  Week 12: number analyzed (Participants) | 55 | 57
  Week 12 | 65.58182 (1.2581561) | 67.42105 (1.3020967)

4. Secondary Outcome: Screen for Child Anxiety Related Disorders
Description: The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item, dual-informant measure of pediatric anxiety symptoms; we use the mean of the parent and child ratings. The questionnaire consists of five subscales assessing symptoms of generalized anxiety, social anxiety, separation anxiety, panic, and school refusal. Items are rated on a scale from 0 to 2; the overall score range is 0 to 82. Higher scores reflect greater levels of anxiety.
Time Frame: Weeks 3, 8, and 12
Population: The analyses included participants who were randomized to either arm of the study and had data available for analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Intervention | Control Intervention
Number analyzed (Participants) | 59 | 61
units on a scale
  Week 3 | 30.08051 (1.288642) | 30.28443 (1.579966)
  Week 8: number analyzed (Participants) | 51 | 58
  Week 8 | 26.29412 (1.402873) | 28.40000 (1.504715)
  Week 12: number analyzed (Participants) | 53 | 56
  Week 12 | 24.49434 (1.381877) | 25.71429 (1.592165)

5. Secondary Outcome: State-Trait Anxiety Inventory for Children
Description: The level of anxiety was assessed using the State-Trait Anxiety Inventory for Children (STAI-C). STAI-C is a 20-item self-report measure of trait anxiety. Items are rated on a scale from 1 to 3; the overall score range is 20-60. Higher scores reflect greater levels of anxiety. STAI-C score was measured at different time points during the study.
Time Frame: Weeks 3, 8, and 12
Population: The analyses included participants who were randomized to either arm of the study and had data available for analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Intervention | Control Intervention
Number analyzed (Participants) | 56 | 62
units on a scale
  Week 3: number analyzed (Participants) | 56 | 59
  Week 3 | 39.58929 (1.029997) | 38.64407 (1.222658)
  Week 8: number analyzed (Participants) | 53 | 62
  Week 8 | 38.94340 (1.090404) | 38.35484 (1.089612)
  Week 12: number analyzed (Participants) | 56 | 56
  Week 12 | 36.92857 (1.011254) | 36.55357 (1.162431)

6. Secondary Outcome: Self-Efficacy Questionnaire
Description: The Self-Efficacy Questionnaire (SEQ-C) is a 24-item self-report measure of self-efficacy in youth. The questionnaire is made up of three subscales assessing social self-efficacy, academic self-efficacy, and emotional self-efficacy. Items are rated on a scale from 1 to 5; the overall score range is 24-120. Higher scores reflect higher levels of self-efficacy.
Time Frame: Pre-Treatment Screening, Weeks 3, and 12
Population: The analyses included participants who were randomized to either arm of the study and had data available for analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Intervention | Control Intervention
Number analyzed (Participants) | 56 | 56
units on a scale
  Pre-Treatment: number analyzed (Participants) | 40 | 39
  Pre-Treatment | 69.65 (2.116646) | 77.61538 (2.124853)
  Week 3: number analyzed (Participants) | 55 | 56
  Week 3 | 71.76364 (1.770876) | 75.21429 (2.024158)
  Week 12: number analyzed (Participants) | 56 | 54
  Week 12 | 77.57143 (1.897342) | 78.07407 (1.964011)

ADVERSE EVENTS:
Time Frame: Up to 9 months
Arm/Group | Active Intervention | Control Intervention
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/62
Serious Adverse Events (participants affected / at risk) | 3/59 | 1/62
Other Adverse Events (participants affected / at risk) | 7/59 | 7/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Intervention (N=59) | Control Intervention (N=62)
Intentional self-injury (Psychiatric disorders) | 1 | 0
Self-injurious ideation (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Intervention (N=59) | Control Intervention (N=62)
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 1 | 1
Concussion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 3
Sedation (Nervous system disorders) | 0 | 1
Blunted affect (Psychiatric disorders) | 1 | 1
Dermatillomania (Psychiatric disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT03283930/Prot_SAP_000.pdf